CLINICAL TRIAL: NCT04861272
Title: RISK PERCEPTION ASSOCIATED WITH COVID-19 PANDEMIC AMONG ANESTHETISTS: A Cross-Sectional Study
Brief Title: Risk Perception Associated With Covid-19 Among Anesthetists
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, SALAH EL-TALLAWY, Professor and Consultant - Anesthesia and Pain Management, King Saud University
Other Study IDs: IRB approval No. E-20-4975
Record Dates: First submitted 2021-04-25; First posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Cross Sectional Hospital Based Study
Keywords: COVID-19 pandemic, Anesthetists, Psychological stress, Anxiety, Depression, PTSD
MeSH Terms: conditions — COVID-19; Stress, Psychological; Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Survey — Online survey

SUMMARY:
Since the outbreak of the COVID-19 pandemic, the anesthesiologists are involved in the riskiest interventions e.g. airway management, endotracheal intubation, and resuscitation. So, they are subjected to a higher risk of infection compared to many other medical specialties. As a result, they are more subjected to psychological stresses. This study aimed to assess the level of stress associated with the COVID-19 pandemic among anesthesiologists.

DETAILED DESCRIPTION:
This is a cross-sectional, hospital-based survey conducted using an online questionnaire after getting IRB approval. The primary outcomes are to evaluate the prevalence of anxiety, depression, and post-traumatic stress disorder (PTSD) among anesthesiologists working in Saudi Arabia. The secondary outcomes include the association of the socio-demographic and occupational characteristics with mental health in the study sample. The survey sent to the target participants using a web-based software platform (https://www.surveymonkey.com/r/ZJ98BTJ) though the Saudi Society of Anesthesia. The study sample included anesthetists and their allied health care providers (nurses and technicians) involved in the management of COVID-19 patients. Data were analyzed using SPSS version 21. Descriptive analyses were conducted, and the ranked data for each level for symptoms of depression, anxiety, and PTSD were presented as numbers and percentages. Multi-variable logistic regression analysis was used to explore potential influence factors on the outcomes. P-values of less than 0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* The survey included anesthesia physicians, anesthesia technicians and nurses, and those involved in the management of COVID-19 infected patients in the OR, ICU, or ER.

Exclusion Criteria:

* The exclusion criteria include age < 18 or > 60 years, incomplete data, or those who were outside Saudi Arabia during the time of the COVID-19 pandemic.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Participants' demographic variables such as gender, age, years of experience, educational degree, position at the hospital, unit of work and hospital type.
  * Outcome variables: The prevalence of Anxiety, Depression and Posttraumatic Stress Disorder (PTSD)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-05-05 (Estimated); Study Completion 2021-05-15 (Estimated)

PRIMARY OUTCOMES:
- The prevalence of Anxiety, Depression, and Posttraumatic Stress Disorder (PTSD) among anesthesiologists during COVID-19 pandemic. | 2 weeks
  Online survey

SECONDARY OUTCOMES:
- Comparison of the prevalence of anxiety, depression, and level of stress among different groups e.g. males # females, different occupations, single # married, young, middle-aged # geriatrics | 2 weeks
  Online survey

CONTACTS AND LOCATIONS:
Overall Officials: SALAH N. EL-TALLAWY, MD, Principal Investigator — KING SAUD UNIVERSITY, Riyadh, Saudi Arabia
Locations (1):
- Salah N. El-Tallawy, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No